CLINICAL TRIAL: NCT02455505
Title: Identifying Family Members in Need of Support While Caregiving and After Loss
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Calvary Hospital, Bronx, NY (Other); The New School for Social Research (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 15-095
Record Dates: First submitted 2015-05-22; First posted 2015-05-28 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Advanced Cancer
Keywords: Cancer Care and Bereavement; Supportive Care; 15-095

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Risk Screening tool & Cognitive Interview
  Interventions: Behavioral: background questionnaire; Behavioral: bereavement risk screening tool

INTERVENTIONS:
Behavioral: background questionnaire
Behavioral: bereavement risk screening tool

SUMMARY:
This screening tool will be used to identify significant relations of patients with advanced medical illness or serious hospitalization and family individuals who lost their loved one and who could use professional support in the future. We are interested in enrolling family members or close friends of patients with advanced medical illness as well as family members or close friends who have lost a loved one. Some screening tools to identify family members who might need support do exist, but the investigators are hoping to develop one that is brief and easier for healthcare providers to use. The information learned in this study will help us refine the screening tool. Family member input will be essential in the development of this screening tool.

ELIGIBILITY:
Inclusion Criteria:

* As per self-report, 21 years or older
* As per self-report, has a domestic partner or spouse, child (minor or adult), sibling (sister or brother), parent or close friend diagnosed with any advanced medical illness or who was recently (2 months) or is currently hospitalized for life-threatening injuries or conditions related to a traumatic incident (e.g., car accident, overdose, assault) OR
* As per self-report, experienced the recent (within 2 months to 3 years) death of a domestic partner or spouse, child (minor or adult), sibling, parent or close friend.
* Responds "yes" to the question "Can you understand spoken and written English?
* Agrees to be audio-taped during the cognitive interview [Waves 1 and 2 only] * For Part 2 only: In the event that the patient dies prior to a consenting pre-loss family member completing the study questionnaires, the family member will be eligible for participation in the post-loss group after at least 2 months have passed after the loss

Exclusion Criteria:

* Significant psychiatric or cognitive disturbance sufficient, in the investigators' judgment, to preclude the completion of the assessment measures or informed consent (i.e., acute psychiatric or neurological symptoms which require individual treatment)
* Another family member (parent, domestic partner or spouse, sibling, or adult child) has been enrolled in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from MSK and Calvary Hospital locations (The Bronx, Brooklyn, and Manhattan), which provides hospice and bereavement services to patients suffering from advanced cancer and their families.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2015-05; Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
to refine the bereavement risk screening tool and its items based on respondent feedback. | 1 year
  we will obtain family member input on the pre- and post-loss versions of the screening tool; we will obtain input from a separate sample of family members on a revised version of the screening tool that incorporates feedback

CONTACTS AND LOCATIONS:
Overall Officials: William Rosa, PhD, MBE, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Calvary Hospital, The Bronx, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/